CLINICAL TRIAL: NCT04782258
Title: A Phase 3b Multicenter Open-label Trial of the Safety, Tolerability, and Efficacy of Tolvaptan in Infants and Children 28 Days to Less Than 18 Years of Age With Autosomal Recessive Polycystic Kidney Disease (ARPKD)
Brief Title: A Study to See Iftolvaptan is Safe in Infants and Children Who at Enrollment Are 28 Days to Less Than 18 Years Old withAutosomal Recessive Polycystic Kidney Disease (ARPKD)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 156-201-00307; 2020-005992-10 (EudraCT Number)
Record Dates: First submitted 2021-02-19; First posted 2021-03-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Autosomal Recessive Polycystic Kidney (ARPKD)
Keywords: ARPKD; TOLVAPTAN; Polycystic Kidney Disease; Autosomal Recessive Polycystic Kidney Disease; Adolescent; Renal Cysts; Oligohydramnios; Anhydramnios
MeSH Terms: conditions — Polycystic Kidney, Autosomal Recessive; Polycystic Kidney Diseases; Oligohydramnios | interventions — Tolvaptan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tolvaptan Suspension (Experimental): Tolvaptan suspension will be administered orally or via feeding/nasogastric tube at doses of 0.15 mg/kg once daily in the AM, 0.30 mg/kg once daily in the AM, 0.5 mg/kg once daily in the AM, 0.75 mg/kg split dose (0.5 mg/kg AM and 0.25 mg/kg 8 hours later), and 1 mg/kg split dose (0.67 mg/kg AM and 0.33 mg/kg 8 hours later) based on age. Treatment duration is 18 months.
  Interventions: Drug: Tolvaptan Suspension
- Tolvaptan Tablets (Experimental): Tolvaptan tablets will be administered orally as split-dose regimens (15/7.5 mg, 30/15 mg, and 45/15 mg) upon awakening and 8 hours later (twice daily) based on weight if able to swallow tablets. Treatment duration is 18 months.
  Interventions: Drug: Tolvaptan Tablets

INTERVENTIONS:
Drug: Tolvaptan Suspension — Syrup
  Arms: Tolvaptan Suspension
Drug: Tolvaptan Tablets — Tolvaptan (OPC-41061) Tolvaptan tablets will be administered orally as split-dose regimens (15/7.5 mg, 30/15 mg, and 45/15 mg) upon awakening and 8 hours later (twice daily) based on weight if able to swallow tablets.
  Arms: Tolvaptan Tablets

SUMMARY:
To evaluate the safety of tolvaptan in pediatric subjects with ARPKD

DETAILED DESCRIPTION:
This study is a multinational, multicenter, open-label, non-randomized trial. The study consist of three periods: Screening Period, Treatment period and Follow-up period.

Tolvaptan has been demonstrated to delay the decline of kidney function in adults with rapidly progressing ADPKD (CKD stages 1 to 4), a closely related indication to ARPKD, as measured by estimated glomerular filtration rate (eGFR) and Total Kidney Volume (TKV).

Participants in this study will be assigned to tolvaptan and followed for 18 months over the course of the study.

The overall trial duration is expected to be approximately 3.5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 28 days and less than 18 years of age, with clinical features that are consistent with a diagnosis of ARPKD.
2. Ability for parent/legal guardian to provide written, informed consent prior to initiation of any trial-related procedures, and ability, in the opinion of the principal investigator, to comply with all the requirements of the trial. Ability to provide written informed assent from all subjects old enough per local laws to provide assent.

Exclusion Criteria:

1. Premature birth (≤ 32 weeks gestational age) for infants 28 days to < 12 weeks of age.
2. Anuria or RRT defined as intermittent or continuous hemodialysis, peritoneal dialysis, hemofiltration, hemodiafiltration or history of kidney transplantation.
3. Evidence of syndromic conditions associated with renal cysts (other than ARPKD).
4. Abnormal liver function tests including ALT and AST, > 1.2 × ULN (upper limit of normal).
5. Has splenomegaly or portal hypertension (HTN).
6. Parents with renal cystic disease.
7. Receiving chronic diuretic that could not be adjusted after tolvaptan initiation.
8. Cannot be monitored for fluid balance.
9. Has or at risk of having sodium and potassium electrolyte imbalances, as determined by the investigator.
10. Has or at risk of having significant hypovolemia as determined by investigator.
11. Clinically significant anemia, as determined by investigator.
12. Platelets < 50000 µL.
13. Severe systolic dysfunction defined as ejection fraction < 14%.
14. Serum sodium levels < 130 mmol/L or >145 mmol/L.
15. Taking any other experimental medications.
16. Require ventilator support.
17. Taking medications known to induce CYP3A4 (CYP = Cytochrome P).
18. Having an infection including viral that would require therapy disruptive to IMP dosing.
19. Females who are breast-feeding or who have a positive pregnancy test result prior to receiving IMP.
20. Subjects with a history of substance abuse (within the last 6 months).
21. Subjects who have bladder dysfunction and/or difficulty voiding.
22. Subjects taking a vasopressin agonist (eg, desmopressin).
23. Subjects with a history of persistent noncompliance with antihypertensive or other important medical therapy.
24. Subjects taking medications or having concomitant illnesses likely to confound endpoint assessments, including taking approved (ie, marketed) therapies for the purpose of affecting PKD cysts such as tolvaptan, vasopressin antagonists, anti-sense ribonucleic acid (RNA) therapies, rapamycin, sirolimus, everolimus, or somatostatin analogs (ie, octreotide, sandostatin).
25. Received or are scheduled to receive a liver transplant.
26. History of cholangitis within the last 6 months.
27. Has findings consistent with clinically significant portal hypertension (eg, varices, variceal bleeding, hypersplenism indicated by thrombocytopenia).

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-08-14 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs) | Enrollment up to 7 days post last dose

SECONDARY OUTCOMES:
Annual rate of change of eGFR (by Schwartz formula) from baseline to post-treatment after 18 months of treatment | From Enrollment to 18 months
Change from baseline of eGFR (by Schwartz formula) while on treatment at Months 1, 6, 12, and 18 | 1 month, 6 months, 12 months, and 18 months
The percentage of subjects that will receive renal replacement therapy (RRT) by 18 months. | From Enrollment to 18 months
The amount of time between enrollment and 18 months that a subject requires renal replacement therapy (RRT). | From enrollment to 18 months

CONTACTS AND LOCATIONS:
Locations (23):
- United States (12):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine - Ann & Robert H. Lurie Children's Hospital of Chicago - Neonatology, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Children's Hospital - New Orleans, New Orleans, Louisiana
  - Johns Hopkins Pediatric Specialty Clinic, Baltimore, Maryland
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Primary Children's Hospital, Salt Lake City, Utah
- Belgium (3):
  - Université Catholique De Louvain And Cliniques St Luc, Brussels, Brussels Capital
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams Brabant
- Universitätsklinikum Köln, Cologne, North Rhine-Westphalia, Germany
- Poland (2):
  - Instytut "Pomnik - Centrum Zdrowia Dziecka", Warsaw, Masovian Voivodeship
  - Uniwersytecki Dzieciecy Szpital Kliniczny im. L. Zamenhofa, Bialystok
- Spain (4):
  - Universitat de Barcelona - Hospital Sant Joan de Deu Barcelona (HSJDB), Esplugues de Llobregat, Barcelona
  - Hospital Universitari Parc Tauli, Sabadell, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Universitario Virgen del Rocío Avenida Manuel Siurot, Seville
- Great Ormond Street Hospital for Children NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Otsuka Clinical Trials Website — https://trials.otsuka-us.com/